CLINICAL TRIAL: NCT01929005
Title: Integrated Inpatient/Outpatient Care for Patients at High Risk of Hospitalization
Brief Title: Comprehensive Care Physician: Integrated Inpatient and Outpatient Care for Patients at High Risk of Hospitalization
Acronym: CCP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University HealthSystem Consortium (Other); University of Illinois at Chicago (Other); Rush University Medical Center (Other); Northwestern University (Other); Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB12-1440; FP050658-01-PR (Other Grant/Funding Number: Centers for Medicare and Medicaid Services)
Record Dates: First submitted 2013-06-29; First posted 2013-08-27 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Medicare Patients; High Risk of Hospitalizations
Keywords: Comprehensive care; Medicare; Cost-sharing; Quality of care
MeSH Terms: interventions — Comprehensive Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): If patients are randomized to standard of care, they are not assigned to a Comprehensive Care Physician. They are asked to continue receiving their care as they normally would.
- Comprehensive Care (Experimental): Patients randomized to the Comprehensive Care group are assigned to a Comprehensive Care physician and are asked to see their assigned CCP for their primary care. The patients will receive their care by the CCP in the outpatient clinic and also if they were to be hospitalized.
  Interventions: Other: Comprehensive Care

INTERVENTIONS:
Other: Comprehensive Care — Patients will receive comprehensive medical care from their CCP in clinic and the hospital. For most patients, the ambulatory care provided by the CCP will be in our onsite medicine clinic, but for some patients with subspecialty needs the CCP may be a specialist who will care for the patient in a nearby ambulatory setting (e.g., nursing home, dialysis facility). The CCPs will also supervise the nurses, pharmacists, social workers, and others who are part of the multi-disciplinary care team. Daytime inpatient care will be provided by CCPs in conjunction with our inpatient advanced practice nurses (APNs). These APNs now work with our hospitalists, so they are experienced providing hospital care.
  Arms: Comprehensive Care

SUMMARY:
The investigators propose an innovative new model of care in which patients identified to be at high risk of hospitalization are offered care by a physician who will direct their care both in the hospital and in clinic but is able to do so because they see patients only at high risk of hospitalization. This allows these physicians to have a panel of patients that is small enough that they can provide them with continuing ambulatory care but sick enough for those physicians to have enough of their patients hospitalized at any time to justify having the physician spend several hours each morning seeing those patients in the hospital, making the model economically viable and clinically valuable for the patient. The investigators estimate that each of the 5 physicians the investigators propose to establish in this model will serve a panel of about 200 patients in steady state with an average of 10 days of expected hospitalization and $75,000 each in Medicare spending per year, totaling $75 million annually. The investigators estimate that a 1% reduction in costs for these patients will be more than enough to cover the ongoing costs of the model the investigators propose; this is because the investigators' program reorganizes care rather than adding new forms of care.

DETAILED DESCRIPTION:
The investigators' project has 5 aims:

Aim 1: To implement an innovative Comprehensive Care Physician (CCP) Model of multi-disciplinary team-based care at the University of Chicago Medical Center (UCMC) in which care for patients at high risk of hospitalization is led by CCPs who focus their practices on patients at high risk of hospitalization so that they can personally care for these patients both in clinic and in the hospital, with savings to Medicare shared with the AMC.

As noted above and supported by theory and data below, the key justification for this goal is based on the value of the doctor-patient relationship. Building on 15 years experience developing our hospitalist program (IRB protocol 9967) from 2 to 30 clinicians, the investigators provide detailed plans to efficiently implement the investigators' model to improve care within 6 months. To incentivize and assess cost-savings, the investigators propose:

Aim 2: Among patients who meet clinical eligibility criteria for the CCP model and express willingness to receive care in the model, to assess the utilization and quality of health care, health outcomes, and cost of care of patients randomly assigned to be offered CCP care compared to patients randomly assigned not to be offered CCP care.

Evaluation is important in the investigators' project both to ensure that the investigators meet the triple-aim and because assessment of cost savings is needed to implement the shared savings model that the investigators think is important to incentivize cost savings. The investigators recognize that the use of randomization to assess out-comes cannot be the basis for a long-term payment model in Medicare but select this approach to evaluation because the investigators think it will provide the most accurate estimate of the effects of the program. Assuming capitated payments to Accountable Care Organizations (ACOs) become a major payment approach for Medicare, cost savings from CCPs would create sustainable incentives for their use. CCPs might also work well in ACOs because selection of high risk patients into a CCP program might not be a concern if those patient came from within the ACO's covered population. Sustained incentives to use CCPs could also exist if high-risk persons selected into ACOs with CCPs, but risk adjustment was adequate. Shared savings programs with adequate risk adjustment would produce similar incentives. To address dissemination and risk adjustment, the investigators propose:

Aim 3: To use data collected by UHC from 4 Chicago-area AMCs with linked Medicare data to support evaluation and potential local and national dissemination of the CCP model

UHC (previously University HealthSystem Consortium) includes over 100 AMCs nation-wide and has exceptional data on hospital resource use to support risk-adjustment. UHC also houses laboratory and Medicare data to enhance risk-adjustment and outcomes assessment. The investigators will use this data to inform potential local dissemination and testing of our model by helping the other participating Chicago-area AMCs identify the segments of their patient populations that are frequently admitted enough to be suitable for the CCP model. If the model is successful at UCMC, and perhaps in later local dissemination and evaluation, UHC's national scope creates opportunities for dissemination of the investigators' work to almost all US AMCs. The risk-adjustment data will also allow us to evaluate alternative strategies to assess program savings to estimate shared savings that do not require randomization. Thus the investigators propose:

Aim 4: To compare the results obtained in Aim 2 to three alternative assessment strategies that: 1) compare patients in UCMC treated in the CCP model to patients in UCMC who meet CCP clinical eligibility criteria but receive usual care, 2) compare patients in UCMC who meet CCP clinical eligibility criteria to historical patients in UCMC who met CCP clinical eligibility criteria, 3) compare patients in UCMC eligible for the CCP model to current patients in 4 other Chicago-area AMCs who meet CCP clinical eligibility criteria.

The investigators propose to evaluate these alternative approaches for selection of a control group because the investigators think they might be feasible approaches to estimate savings in a shared-savings model and because they differ in potential threats to validity (e.g., 1 must address patient selection into the intervention and 2 must address time trends in costs), outcomes assessment (patient outcomes will be harder to assess in 2 and 3), and generalizability (1 requires local patients treated outside the model and 2 requires historical data, which becomes less relevant over time). All models will be adjusted with the CMS-Hierarchical Condition Category (HCC) risk adjustment model for our base analysis but the investigators will also explore other approaches to risk adjustment, such as using prior year total Medicare expenditures and patient-reported variables as risk adjusters. The investigators propose to use our randomized control group for our shared savings incentive, but to work with CMMI in our cooperative agreement to assess how these control groups and approaches to risk adjustment could be used in shared savings incentives. Patient-reported outcomes will be assessed from enrolled subjects. Finally, since workforce development is key to implementing and disseminating this model, the investigators propose:

Aim 5: To develop skills of a multidisciplinary team of providers to execute the CCP model, and expose medical students, residents and fellows, and other health professions trainees to the model.

Because the investigators are an AMC with a rich pipeline of health professions trainees and excellent record of training national leaders, the investigators are excellently situated to train clinicians in the investigators' model who have the potential to help disseminate its core principles both locally and nationally.

ELIGIBILITY:
Inclusion Criteria:

* Medicare recipients and were hospitalized at least one time in the past year

Exclusion Criteria:

* Non-Medicare recipients and/or were not hospitalized in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2008 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | Every 3 months after patient enrollment up to 3 years
  patient satisfaction measured by Consumer Assessment of Health Plans (CAHPs) instrument
Total Cost of Care | Cumulative costs after enrollment up to 3 years
  Total cost of care will be measured using Medicare claims data obtained from RESDAC to examine all care that charged to Medicare, including use of acute care hospitals, physician services, SNF, home health, hospice, etc., and Part D. We will also seek to link to data from Illinois Medicaid for our dual eligibles.

SECONDARY OUTCOMES:
Patient outcomes | Every 3 months after enrollment up to 3 years
  Patient outcomes will be measured by quarterly assessment by phone of health status using the SF-12, limitations of activities of daily living (ADLs) and instrumental ADLs (IADLs) and patient satisfaction (e.g., Consumer Assessment of Health Plans (CAHPs) instrument).
Care utilization | Cumulative utilization from patient enrollment up to 3 years
  Following Donabedian's framework, we will first assess the extent to which care is structured with integrity to the CCP model using a primary measure of what fraction of a patient's clinic and hospital encounters are provided by their CCP. Care utilization will be measured using Medicare claims data obtained from RESDAC to examine all care that charged to Medicare, including use of acute care hospitals, physician services, SNF, home health, hospice, etc., and Part D. We are experienced working with these raw claim files for research. We will also link to data from Illinois Medicaid for our dual eligibles. For utilization in the hospital (e.g., ICU days or ICU days in terminal hospitalization), we will use UHC data.
Doctor-patient relationship | Every 3 months after enrollment up to 3 years
  Given the central role of the quality of the doctor-patient relationship on our conceptual model of care, we will administer the Primary Care Assessment Survey (discussed above) quarterly.
Mortality | Cumulative after enrollment up to 3 years
  Mortality will be assessed by report of key contacts and confirmed using death records.

OTHER OUTCOMES:
Provider outcomes | Every 6 months beginning at the start of data collection up to 3 years
  Provider outcomes are also important. We have surveyed attending physician about job satisfaction for 15 years with multiple domains including satisfaction with ability to provide high quality care, efficient care, relationships with patients, relationships with providers, etc., and will continue these annually for all our attendings and for our CCPs. However, with only 5 CCPs, qualitative reports will be most valuable so we will interview them quarterly, transcribing comments for formal qualitative analysis. Given the tiny number of CCPs, all CCPs will be allowed to review resulting manuscripts before submission and redact elements as they feel appropriate, either out of personal interest or belief that a clinical reference might be identified with a specific patient.

CONTACTS AND LOCATIONS:
Overall Officials: David Meltzer, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No